CLINICAL TRIAL: NCT06179979
Title: PET Study With 11 C-PIB to Evaluate Amyloid Protein Deposits in Mild Cognitive Disorder, Alzheimer's Disease and Early Frontotemporal Degeneration.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PET-PIB-1
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET/CT with 11C-PiB — Subjects considered suitable will undergo a clinical and neuropsychological evaluation and a PET/CT study with intravenous administration of 11C-PIB.

SUMMARY:
Preclinical and clinical data have demonstrated the ability of the 11C-PIB tracer to selectively bind accumulations of amyloid protein, a neuropathological marker characteristic of the neurodegenerative pathologies covered by this study.

The validation in larger groups of patients, and the comparison between the different clinical syndromes included in the spectrum, will allow the diagnostic and prognostic potential of the tracer to be evaluated, with important consequences for the clinical management of patients.

In particular, the tracer could play a central role in the clinical management of patients with neurodegenerative diseases and cognitive impairment.

Numerous pharmacological trials are currently underway, worldwide, for the validation of anti-amyloid drugs. In the future we could think about early monitoring with imaging of the effectiveness of the treatment.

T he FDG PET technique can be of great help in obtaining relationships between radiation damage to the brain and possibly neurological and neuropsychological deficits associates.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's diagnosis according to the diagnostic criteria in use.

Exclusion Criteria:

* current or previous treatments with neuroactive drugs;
* pregnancy or breastfeeding.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with neurodegenerative diseases will be included: with mild cognitive disorder, Alzheimer's dementia and early temporal frontal degeneration.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-05-17 (Actual); Primary Completion 2008-07-15 (Actual); Study Completion 2008-07-15 (Actual)

PRIMARY OUTCOMES:
PET/CT with 11C-PiB to characterize amyloid protein deposits in patients with neurodegenerative diseases. | 2 years
  Comparative evaluation of the accumulation of amyloid protein in the various neurodegenerative conditions included with attention to the specificity of the tracer as an element of differential diagnosis.

IPD SHARING:
Plan to Share IPD: No